CLINICAL TRIAL: NCT05185583
Title: A Phase II Proof-of-concept Trial of Methylphenidate in Children With Apraxia of Speech: a Double-blind, Randomised, Placebo-controlled, Cross-over Trial
Brief Title: Methylphenidate in Childhood Apraxia of Speech
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 77169
Record Dates: First submitted 2021-11-29; First posted 2022-01-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Childhood Apraxia of Speech
Keywords: Childhood Apraxia of Speech; Methylphenidate; Ritalin; Developmental Verbal Apraxia; Apraxia, Verbal; Attention Deficit-Hyperactivity Disorder; Central Stimulants; Central Nervous System (CNS) Stimulants; Intelligibility, Speech
MeSH Terms: conditions — Apraxias; Attention Deficit Disorder with Hyperactivity; Speech Intelligibility | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sequence A: Methylphenidate, Placebo (Experimental): Participants will first receive methylphenidate capsules twice daily for four weeks. Doses will be administered four hours apart. The maximum dose is determined based on the participant's weight. After a 2-day washout, participants then receive Placebo (matching methylphenidate capsules) twice daily for four weeks.
  Interventions: Drug: Methylphenidate Hydrochloride; Drug: Placebo
- Sequence B: Placebo, Methylphenidate (Experimental): Participants will first receive Placebo capsules twice daily for four weeks. Doses will be administered four hours apart. After a 2-day washout, participants then receive methylphenidate capsules (matching Placebo capsules) twice daily for four weeks. The maximum dose is determined based on the participant's weight.
  Interventions: Drug: Methylphenidate Hydrochloride; Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate Hydrochloride — Participants will receive twice daily doses of Methylphenidate Hydrochloride four hours apart. There will be three dosage schedules, determined based on three weight ranges (20-30kg; 30-40kg; ≥40kg). For children weighing 20-30kg, the maximum daily dose will be 20mg. For children weighing 30-40kg, the maximum daily dose will be 30mg. For children weighing ≥40kg, the maximum daily dose will be 40mg.
  Other Names: Ritalin 10
Drug: Placebo — Participants will receive twice daily doses of placebo capsules. Gelatine placebo capsules will contain hypromellose, an inert substance.

SUMMARY:
The purpose of this study is to describe the possible effects of methylphenidate (MPH) on speech intelligibility in children with childhood apraxia of speech (CAS) aged 6-12 years. This outcome will be compared between MPH intake and placebo intake.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, two-period crossover proof-of-concept trial of methylphenidate (MPH) for children with childhood apraxia of speech (CAS). 24 children aged 6 to 12 years with CAS will be recruited. If children pass the screening procedure, which includes a physical exam conducted by a medical officer at the Melbourne Children's Campus, children will be enrolled into the 8 weeks + 2-day trial (includes 2-day washout). Participants will be randomly assigned to sequence A (4 weeks of MPH, followed by 4 weeks of placebo) or sequence B (4 weeks of placebo, followed by 4 weeks of MPH). After 4 weeks in period 1, a two-day washout period will occur before participants crossover to period 2 for 4 weeks. Pre- and post-treatment speech outcomes will be measured. The investigators' primary objective is to provide proof-of-concept that speech intelligibility could demonstrate greater improvements from baseline to 4 weeks following a 4-week period of MPH use compared with placebo in children with CAS. The secondary objectives are to describe feasibility, tolerability and change from baseline in: connected speech intelligibility, quality of language production, speech quality, functional speech intelligibility, phonological working memory, attentional and hyperactive behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Has childhood apraxia of speech
* Aged 6-12 years
* Can perform the speech tasks for the trial (able to speak single words and short sentences)
* English as a first language
* Has adequate hearing
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on their behalf
* Passes the health and medical examination including examination of heart rate and blood pressure for age and weight norms
* Can commit to the time requirements of the trial
* Lives within 250 kilometres of the study site (MCRI)
* Able to swallow a capsule
* Scores 13 or more out of 27 on either the inattention and/or hyperactivity subscales of the SNAP-IV Parent 18-Item Rating Scale, suggesting clinically significant symptoms of inattention and/or hyperactivity

Exclusion Criteria:

* Is unable to commit to the time requirements of the trial (8 weeks + 2 days)
* Has a diagnosis of severe intellectual disability, or other significant neurodevelopmental conditions (e.g., Fragile X, Down Syndrome, etc.)
* Has epilepsy or other seizure disorders
* Is taking medication(s) for another health condition(s) that is known to interfere with MPH
* Has any contraindication to the stimulant (methylphenidate) medication, including severe anxiety, depression, severe Tourette syndrome, glaucoma, psychotic symptoms, hypertension, congenital heart disease, known past or present diagnosed substance abuse or dependence
* Has a score of moderate or high risk of suicidality, assessed with the Columbia Suicidality Severity Rating Scale (C-SSRS)
* Has used psychostimulants within the past 3 months (e.g., Ritalin, Concerta, Focalin)
* Lives more than 250 kilometres from the study site
* Unable to swallow a capsule

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Preschool Speech Intelligibility Measure Score at 4 weeks | Baseline and 4 weeks
  Single word speech intelligibility will be measured using the Preschool Speech Intelligibility Measure (PSIM). Twenty (20) items from the PSIM will be administered at each testing time point. Participants are required to repeat each test word after the researcher. Higher scores are indicative of greater unintelligibility (range 0-80). Mean change from baseline will be reported at the group level.

SECONDARY OUTCOMES:
Change From Baseline in Assessment of the Intelligibility of Dysarthric Speech-II (ASSIDS-II) Score at 4 weeks | Baseline and 4 weeks
  The Assessment of the Intelligibility of Dysarthric Speech-II (ASSIDS-II) will be used to measure sentence level speech intelligibility. Five (5) 5-word sentences will be administered at each assessment time point. A phonemic accuracy score will be calculated by determining the percentage of correct phonemes across the 5 sentences at each timepoint. Mean change from baseline will be reported at the group level.
Number of children at screening who refuse, are eligible, or are ineligible (and reason). | At study recruitment, up to 4 weeks before starting treatment.
  The frequency of children at screening who refuse, are eligible, or are ineligible (and reason).
Number of children who withdraw, discontinue, and/or experience 1 or more protocol violations. | During the 4 week treatment phase.
  Number of children in either sequence A or B who:
  1. withdraw
  2. discontinue the treatment prior to 4 weeks
  3. experience 1 or more protocol violations.
Adherence to dose regimen during each 4 week treatment period | 4 weeks
  Adherence will be determined by calculating the percentage of prescribed doses achieved based on the medication diary entries and reconciling against returned dispensed medication. A participant will be considered adherent during a 4-week period if 80% of the prescribed doses are achieved. Data will be aggregated such that the proportion of children who adhere to the dosing regimen in each 4-week period will be reported.
Parent/caregiver experience of tolerability and utility | Baseline and 4 weeks
  Measured using the investigators' parent/caregiver tolerability and utility survey which is a dedicated electronic Case Report Form. This provides data on caregiver(s)'s views of usability (e.g., "It was convenient to give my child the capsules"), tolerability (e.g., "It was not a burden to participate in this trial") and experience of the trial (Vogel, 2016) (e.g., "I am glad my child participated in this trial"), and whether speech was improved (e.g., "I think the capsule improved my child's speech"). Items will be rated 1-5 where a score of 1 indicates the parent/caregiver strongly disagrees and a score of 5 indicates the parent/caregiver strongly agrees. One item related to school can be rated as 0 if the child is on holidays or in a COVID-19 lockdown for the trial duration. Total scores range from 20-105, where a higher score indicates a greater tolerability/utility of the trial as rated by the parent. Mean change from baseline will be reported at the group level.
Paediatric patient experience of tolerability and utility | Baseline and 4 weeks
  Measured using the investigators' patient tolerability and utility survey which is a dedicated electronic Case Report Form (eCRF). This provides data on participants' views of usability (e.g., "It was easy to take the capsules"), tolerability/burden (e.g., "I had enough energy to play when taking the capsules") and experience of the trial (Vogel, 2016) (e.g., "I would do this trial again"), and whether speech was improved (e.g.,"I think my speech is better after taking the capsules"). Items will be rated 1-5 where a score of 1 indicates the participant strongly disagrees with the statement and a score of 5 indicates the participant strongly agrees. One item related to school can be rated as 0 if the child is on holidays or in a COVID-19 lockdown for the duration of the trial. Total scores range from 20-105, where, a higher score indicates a greater tolerability/utility of the trial as rated by the child participant. Mean change from baseline will be reported at the group level.
Change From Baseline in total number of grammatical features (Language Assessment, Remediation and Screening Procedure; LARSP) at 4 weeks | Baseline and 4 weeks
  Children's conversational speech will be analysed to determine the total number of grammatical features present using the Language Assessment, Remediation and Screening Procedure (LARSP). Mean change from baseline will be reported at the group level.
Change From Baseline in total number of sentences (Language Assessment, Remediation and Screening Procedure; LARSP) at 4 weeks | Baseline and 4 weeks
  Children's conversational speech will be analysed to determine the total number of sentences present using the Language Assessment, Remediation and Screening Procedure (LARSP). Mean change from baseline will be reported at the group level.
Change From Baseline in mean number of sentences per turn (Language Assessment, Remediation and Screening Procedure; LARSP) at 4 weeks | Baseline and 4 weeks
  Children's conversational speech will be analysed to determine the total number of sentences per turn using the Language Assessment, Remediation and Screening Procedure (LARSP). Mean change from baseline will be reported at the group level.
Change From Baseline in mean sentence length (Language Assessment, Remediation and Screening Procedure; LARSP) at 4 weeks | Baseline and 4 weeks
  Children's conversational speech will be analysed to determine the mean sentence length produced using the Language Assessment, Remediation and Screening Procedure (LARSP). Mean change from baseline will be reported at the group level.
Change From Baseline in stage of grammatical development (Language Assessment, Remediation and Screening Procedure; LARSP) at 4 weeks | Baseline and 4 weeks
  Children's conversational speech will be analysed to determine the child's stage of grammatical development, identified using the Language Assessment, Remediation and Screening Procedure (LARSP). Mean change from baseline will be reported at the group level.
Change From Baseline in types of clausal structures used (Language Assessment, Remediation and Screening Procedure; LARSP) at 4 weeks | Baseline and 4 weeks
  Children's conversational speech will be analysed to determine types of clausal structures used by the child, identified using the Language Assessment, Remediation and Screening Procedure (LARSP). Aggregated data will be reported.
Change From Baseline in syllable repetition at 4 weeks | Baseline and 4 weeks
  Syllable repetition will be measured by analysing the average number of syllables produced, average period or duration between consonant-vowel syllable voicing offsets (milliseconds) and variance of the diadochokinetic period (percentage reported). Mean change from baseline will be reported at the group level, and will be compared between Sequence A and Sequence B.
Change From Baseline in Intelligibility in Context Scale Score at 4 weeks | Baseline and 4 weeks
  The Intelligibility in Context Scale (ICS) will measure functional speech intelligibility using parent/caregiver ratings across 7 items, where high scores are indicative of poor intelligibility of speech (range 7-35). Mean change from baseline will be reported at the group level.
Change From Baseline in Children's Non-word Repetition (CNRep) Test Score at 4 weeks | Baseline and 4 weeks
  The Children's Non-word Repetition (CNRep) Test will measure phonological working memory. Ten CNRep items will be administered at each of the four assessment timepoints to control for learning effects. The percentage of correct responses will be calculated by syllable (i.e., 2, 3, 4 and 5 syllable words) and for the total list of words. Mean change from baseline will be reported at the group level.
Change From Baseline in Swanson, Nolan, and Pelham (SNAP-IV) Parent 18-Item Rating Scale (SNAP-IV) Score at 4 weeks | Baseline and 4 weeks
  The Swanson, Nolan, and Pelham (SNAP-IV) Questionnaire is a measure of Attention Deficit Hyperactivity Disorder (ADHD) symptoms using ADHD diagnostic criteria specified in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV). Parent ratings on the Attention and Hyperactivity subscales will be used to measure attention deficit and hyperactivity symptoms. Higher scores indicate greater inattentive and/or hyperactive behaviours. Scores on each subscale range from 0-27. A score below 13 is indicative of symptoms not being clinically significant. A score of 13-17 indicates mild symptoms; a score of 18-22 indicates moderate symptoms and a score of 22-27 indicates severe symptoms. Mean change from baseline will be reported at the group level.

OTHER OUTCOMES:
Change From Baseline in maximum phonation time at 4 weeks | Baseline and 4 weeks
  Maximum phonation time will be measured by determining the maximum length of a continuous vowel phonation on one breath to indicate airflow sufficiency and adequacy of vocal folds closure. Mean change from baseline will be reported at the group level, and will be compared between Sequence A and Sequence B.
Change from Baseline in vowel space of speech at 4 weeks | Baseline and 4 weeks
  Vowel space measurements can provide objective information on formant distribution and act as a proxy for vowel production. Vowel space will be quantified by using the vowel articulation index (see Sapir et al. (2009) for more information). Mean change from baseline will be reported at the group level, and compared between Sequence A and Sequence B.
Change from Baseline in the Mel-frequency cepstral coefficient (MFCC) at 4 weeks | Baseline and 4 weeks
  Mel-frequency cepstral coefficient (MFCC) measures subtle changes in the motion of the articulators (jaw, tongue, lips). The MFCC coefficient represents the vocal tract transfer function, indicating potential problems in the articulators. The MFCC was designed to represent overall stability of individual vocal tract elements. The MFCC parameter is defined as the mean of the standard deviations of the 1st-12th MFCCs. See Fraile et al. (2009) for further description. Mean change from baseline will be reported at the group level, and compared between Sequence A and Sequence B.
Change from Baseline in mean of pause length of speech at 4 weeks | Baseline and 4 weeks
  The mean of pause length of speech measures the average length of silence in a speech sample. The mean of pause length will be analysed by determining the number of silences divided by the total silence duration (msec). Mean change from baseline will be reported at the group level, and will be compared between Sequence A and Sequence B.
Change from Baseline in standard deviation of pauses of speech at 4 weeks | Baseline and 4 weeks
  The standard deviation of pauses of speech measures the variability in pause length. Mean change from baseline will be reported at the group level, and will be compared between Sequence A and Sequence B.
Change from Baseline in percentage of silence at 4 weeks | Baseline and 4 weeks
  The percentage of silence of speech measures the proportion of silence derived from total pause duration divided by total signal time. Mean change from baseline will be reported at the group level, and will be compared between Sequence A and Sequence B.
Change from Baseline in rate of speech at 4 weeks | Baseline and 4 weeks
  The rate of speech is derived from number of syllables spoken per second. The rate of speech will be analysed by determining the number of syllables spoken in a duration of a speech sample. Mean change from baseline will be reported at the group level, and will be compared between Sequence A and Sequence B.
Change from Baseline in pairwise variability index at 4 weeks | Baseline and 4 weeks
  The Pairwise Variability Index (PVI) is a measure of relative vowel duration across adjacent syllables in a word or sentence that is normalised to allow comparison across different speech rates (Vergis et al., 2014). PVI is calculated by determining the difference in duration for two adjacent syllables and then dividing the difference by an average of the two values. Higher PVI values indicate greater contrastiveness, while values close to zero indicate equal stress. Mean change from baseline will be reported at the group level, and will be compared between Sequence A and Sequence B.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Morgan, PhD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Murdoch Children's Research Institute, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the trial will be available six months after publication of the primary outcome. The study protocol may be obtained from the Murdoch Children's Research Institute. Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the trial investigators must see and approve the analysis plan describing how the data will be analyzed, there must be an agreement around appropriate acknowledgment and any additional costs involved must be covered. Should the study investigators be unavailable, this role is delegated to the Murdoch Children's Research Institute. Data will only be shared with a recognized research institute which has approved the proposed analysis plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication of primary outcome
Access Criteria: Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the trial investigators must see and approve the analysis plan describing how the data will be analyzed, there must be an agreement around appropriate acknowledgment and any additional costs involved must be covered.

REFERENCES:
- [Background] Fraile R, Saenz-Lechon N, Godino-Llorente JI, Osma-Ruiz V, Fredouille C. Automatic detection of laryngeal pathologies in records of sustained vowels by means of mel-frequency cepstral coefficient parameters and differentiation of patients by sex. Folia Phoniatr Logop. 2009;61(3):146-52. doi: 10.1159/000219950. Epub 2009 Jul 1. PMID 19571549
- [Background] Sapir S, Ramig LO, Spielman JL, Fox C. Formant centralization ratio: a proposal for a new acoustic measure of dysarthric speech. J Speech Lang Hear Res. 2010 Feb;53(1):114-25. doi: 10.1044/1092-4388(2009/08-0184). Epub 2009 Nov 30. PMID 19948755
- [Background] Vergis, Ballard, K. J., Duffy, J. R., McNeil, M. R., Scholl, D., & Layfield, C. (2014). An acoustic measure of lexical stress differentiates aphasia and aphasia plus apraxia of speech after stroke. Aphasiology, 28(5), 554-575. https://doi.org/10.1080/02687038.2014.889275
- [Background] Vogel, A., Skarrat, J., Castles, J., Synofzik, M. . (2016). Video game-based speech rehabilitation for reducing dysarthria severity in adults with degenerative ataxia. European Journal of Neurology, 23(227).